CLINICAL TRIAL: NCT06939426
Title: Impact of a Short Music Therapy Program on Intra- and Interpersonal Factors of Humanized Care in a Group of Emergency Nursing Staff at the University Hospital Fundación Santa Fe de Bogotá: a Mixed-methods Pilot and Feasibility Study
Brief Title: Music Therapy and Humanization in ED Healthcare Professionals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Mark Ettenberger, Principal Investigator, Music Therapy Service FSFB, Fundación Santa Fe de Bogota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MTEMERGENCY01
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-04

CONDITIONS: Stress; Burnout; Quality of Life (QOL); Music Therapy; Humanization of Care
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music therapy program (Experimental)
  Interventions: Behavioral: Music therapy intervention

INTERVENTIONS:
Behavioral: Music therapy intervention — The intervention protocol is based on four main themes, which are addressed over the course of eight sessions:
  * Self-care
  * Self-recognition and expression of emotions
  * Empathy
  * Teamwork
  Each theme is related to factors from the HUMAS (affection, self-efficacy, emotional understanding, dispositional optimism, and sociability) and/or ProQOL (compassion satisfaction, burnout, and compassion fatigue). A variety of techniques related to the four main methods of music therapy will be used in the sessions: receptive, re-creative, composition, and improvisation.

SUMMARY:
Background: Healthcare professionals in emergency departments frequently experience stressful situations that could jeopardize their mental health, sense of purpose, and ability to empathize with patients, families, and colleagues.

Research question: What is the impact of a short music therapy program on the intra- and interpersonal factors of humanized care among emergency nursing staff at the University Hospital Fundación Santa Fe de Bogotá (FSFB)? Methodology: This research is a mixed-methods pilot and feasibility study. For the quantitative component, we will apply the HUMAS (Healthcare Professional Humanization Scale) and ProQOL (Professional Quality of Life) measure at the start and at the end of the music therapy program. For the qualitative component, focus group interviews will be conducted and analyzed via thematic analysis.

Discussion: This study seeks to support the nursing staff of the FSFB emergency department through an interactive, creative, and participatory music therapy self-care program focused on one of the most important pillars of the institution: the humanization of care.

ELIGIBILITY:
Inclusion Criteria:

* Be a member of the emergency department nursing staff at the FSFB for a minimum of 6 months.
* Be able to commit to participating in eight music therapy sessions over a four-week period.
* Have the minimum reading skills to understand the questionnaires

Exclusion Criteria:

- Staff with untreated mental health disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
HUMAS (Healthcare Professional Humanization Scale) | From enrollment to the end of the music therapy program after one month
  The HUMAS was developed by Pérez-Fuentes et al. and has been validated in Spanish among nursing professionals. It consists of 19 items evaluated on a 5-point Likert scale, with a total score ranging from 0 to 95, with higher scores indicating greater intra- and interpersonal skills that favor the humanization of the service provided. The items are divided into 5 factors: affection; self-efficacy: emotional understanding; disposition to optimism; sociability.

SECONDARY OUTCOMES:
ProQOL (Professional Quality of Life) measure | From enrollment to the end of the music therapy program after one month
  The ProQOL measure is one of the most widely used scales to determine quality of life in health professionals. It consists of 30 items rated retrospectively (over the past month) on a 5-point Likert scale. The scale measures the following factors: compassion satisfaction, burnout, and compassion fatigue. Each factor scores from 0 to 50, with higher scores indicating a greater satisfaction with an individual's work (compassion satisfaction) or higher scores indicating greater experience of fatigue, stress, or emotional exhaustion (compassion fatigue and burnout). The psychometric properties show satisfactory internal consistency and discriminant validity and it has been recently used in nursing teams in emergency units.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Fundación Santa Fe de Bogotá, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request.
Supporting Information: Study Protocol
Time Frame: After publication of the results without restriction of time.